CLINICAL TRIAL: NCT02293954
Title: Pilot Study: Detection of Carcinomas Using 64Cu-Labeled M5A Antibody to Carcinoembryonic Antigen (CEA)
Brief Title: Copper Cu 64 Anti-CEA Monoclonal Antibody M5A PET in Diagnosing Patients With CEA Positive Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14238; NCI-2014-02079 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14238 (Other: City of Hope Medical Center)
Record Dates: First submitted 2014-10-09; First posted 2014-11-19 (Estimated); Results first posted 2023-04-21 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Colon Cancer; Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Gastrointestinal Cancer; Liver and Intrahepatic Biliary Tract Cancer; Lung Cancer; Metastatic Cancer; Pancreatic Cancer; Rectal Cancer; Thyroid Gland Medullary Carcinoma; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms; Gastrointestinal Neoplasms; Carcinoma, Hepatocellular; Lung Neoplasms; Neoplasm Metastasis; Pancreatic Neoplasms; Rectal Neoplasms; Carcinoma, Medullary | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (copper Cu 64 anti-CEA monoclonal antibody M5A PET) (Experimental): Patients receive copper Cu 64 anti-CEA monoclonal antibody M5A IV on day 0 and then undergo PET on day 1 and day 2.
  Interventions: Procedure: radionuclide imaging; Procedure: positron emission tomography; Other: laboratory biomarker analysis; Other: pharmacological study; Drug: Cu 64 anti-CEA monoclonal antibody M5A IV

INTERVENTIONS:
Procedure: radionuclide imaging — Given copper Cu 64 anti-CEA monoclonal antibody M5A IV
  Other Names: radionuclide scanning
Procedure: positron emission tomography — Undergo PET
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Drug: Cu 64 anti-CEA monoclonal antibody M5A IV — Cu 64 anti-CEA monoclonal antibody M5A IV

SUMMARY:
This pilot clinical trial studies copper Cu 64 anti-carcinoembryonic antigen (CEA) monoclonal antibody M5A positron emission tomography (PET) in diagnosing patients with CEA positive cancer. Diagnostic procedures, such as copper Cu 64 anti-CEA monoclonal antibody M5A PET, may help find and diagnose CEA positive cancer that may not be detected by standard diagnostic methods.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the ability of 64Cu labeled M5A antibody (copper Cu 64 anti-CEA monoclonal antibody M5A) to localize CEA positive cancers (such as gastrointestinal, lung, medullary thyroid and breast cancers), as determined by PET imaging.

SECONDARY OBJECTIVES:

I. To characterize the frequency of titer of the human anti-human antibody (HAHA) response to 64Cu labeled M5A antibody.

II. To determine the safety of administration of 64Cu labeled M5A antibody.

OUTLINE:

Patients receive copper Cu 64 anti-CEA monoclonal antibody M5A intravenously (IV) on day 0 and then undergo PET on day 1 and day 2.

After completion of study, patients are followed up at 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed primary or metastatic cancer; if biopsies were performed at an outside facility, the histology must be reviewed and confirmed by the Department of Pathology at the City of Hope
* Patients must have tumors that produce CEA as documented by a current or past history of an elevated serum CEA above the institutional limit of normal, or by immunohistochemical methods; NOTE: Patients with colorectal cancer are exempt from this requirement since > 95% are CEA positive
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Patients must have a known site of disease; please note, for patients undergoing neoadjuvant therapy, this requirement must be met retrospectively prior to the start of neoadjuvant therapy; patients who are in radiological/clinical remission after neoadjuvant therapy, prior to infusion of radiolabeled antibody, are still eligible
* Although not mandated by the protocol, the results of the CT scan and labs (complete blood count [CBC], comprehensive metabolic panel [CMP]) that are performed as part of the standard work up should be available and should have been done within 2 months prior to study entry
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Prior therapy (chemotherapy, immunotherapy, radiotherapy) must be completed at least 2 weeks prior to infusion of radiolabeled antibody

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to copper Cu 64 anti-CEA monoclonal antibody M5A (64Cu-M5A)
* Patients must not have received prior chemotherapy or radiation for >= 2 weeks before study enrollment
* Pregnant women are excluded from this study; breastfeeding should be discontinued is the mother is treated with 54Cu-m5A
* Any patient who has had exposure to mouse or chimeric (human/mouse) immunoglobulin and has antibody to the M5A
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2022-03-06 (Actual); Study Completion 2026-08-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wong, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Wong JYC, Yamauchi DM, Adhikarla V, Simpson J, Frankel PH, Fong Y, Melstrom KA, Chen YJ, Salehian BD, Woo Y, Dandapani SV, Colcher DM, Poku EK, Yazaki PJ, Wu AM, Shively JE. First-In-Human Pilot PET Immunoimaging Study of 64Cu-Anti-Carcinoembryonic Antigen Monoclonal Antibody (hT84.66-M5A) in Patients with Carcinoembryonic Antigen-Producing Cancers. Cancer Biother Radiopharm. 2023 Feb;38(1):26-37. doi: 10.1089/cbr.2022.0028. Epub 2022 Sep 26. PMID 36154291

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (Copper Cu 64 Anti-CEA Monoclonal Antibody M5A PET): Patients receive 15 mCi/5 mg copper Cu 64 anti-CEA monoclonal antibody M5A IV on day 0 and then undergo PET on day 1 and day 2.
  radionuclide imaging: Given copper Cu 64 anti-CEA monoclonal antibody M5A IV
  positron emission tomography: Undergo PET
  Cu 64 anti-CEA monoclonal antibody M5A IV: Cu 64 anti-CEA monoclonal antibody M5A IV
Period: Overall Study
Arm/Group | Diagnostic (Copper Cu 64 Anti-CEA Monoclonal Antibody M5A PET)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Copper Cu 64 Anti-CEA Monoclonal Antibody M5A PET)
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 57 [21 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4
  Hispanic | 6
  Non-Hispanic White | 10
Region of Enrollment [Number; unit: participants]
  United States | 20
Tumor Stage @ Diagnosis [Count of Participants; unit: Participants] — Stage I, Stage II, and Stage III - Cancer is present. The higher the number, the larger the cancer tumor and the more it has spread into nearby tissues.
  Stage IV - The cancer has spread to distant parts of the body.
  Participants
    I | 1
    II | 1
    III | 5
    IV | 11
    Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Tumor Uptake of 64Cu-DOTA-hT4.66-M5A at Day 1
Description: Tumor uptake measured by SUVmax of 64Cu-DOTA-hT4.66-M5A at day1 for hottest lesion from each patient. For tumors of at least 2 cm in diameter SUV (=tumor activity concentration/injected activity per unit body weight).
Time Frame: At day 1
Measure: Median (Standard Deviation); unit: SUVmax (g/mL)
Arm/Group | Diagnostic (Copper Cu 64 Anti-CEA Monoclonal Antibody M5A PET)
Number analyzed (Participants) | 20
SUVmax (g/mL) | 22.0 (16.9)

2. Primary Outcome: Tumor Uptake of 64Cu-DOTA-hT4.66-M5A at Day 2
Description: Tumor uptake measured by SUVmax of 64Cu-DOTA-hT4.66-M5A at day 2 for hottest lesion from each patient. For tumors of at least 2 cm in diameter SUV (=tumor activity concentration/injected activity per unit body weight).
Time Frame: At day 2
Measure: Mean (Standard Deviation); unit: SUVmax (g/mL)
Arm/Group | Diagnostic (Copper Cu 64 Anti-CEA Monoclonal Antibody M5A PET)
Number analyzed (Participants) | 20
SUVmax (g/mL) | 30.7 (24.4)

3. Secondary Outcome: Number of Participants With Human Anti-human Antibody (HAHA) Positive Response to 64Cu Labeled M5A Antibody
Description: Approximately 5 ml (1 teaspoon) of blood in a red top tube will be drawn at 1 month post study drug infusion and 3 months post study drug infusion. Response at either 1 or 3 months post study drug infusion constitutes a positive response.
Time Frame: At 1 and 3 months post study drug infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Copper Cu 64 Anti-CEA Monoclonal Antibody M5A PET)
Number analyzed (Participants) | 20
Participants | 1

4. Secondary Outcome: The Average Increase of Tumor-to-blood (T:B) Ratio From Day 1 to Day 2
Description: Scan results were compared to known sites of disease as defined by sites identified on CT scans, MRI scans, FDG PET scans, or sites identified at surgery that were histologically positive for cancer. The 64Cu SUVs on both day 1 and 2 scans were evaluated in tumors and selected nontumor organs and tissues (blood pool, liver, spleen, and kidney). Tumor uptake was measured in terms of SUVmax values, while organ uptake to assess biodistribution was measured in terms of SUVmean values. Ratios of tumor-to-blood activity concentration (T:B) were calculated as the ratio of tumor SUVmax to average SUV (SUVmean) measured in the blood pool.
Time Frame: At day 1 and day 2
Measure: Mean (Standard Deviation); unit: T:B
Arm/Group | Diagnostic (Copper Cu 64 Anti-CEA Monoclonal Antibody M5A PET)
Number analyzed (Participants) | 20
T:B
  Day 1 | 3.3 (2.7)
  Day 2 | 6.5 (4.9)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of initial treatment until 30 days post discontinuation of treatment.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Diagnostic (Copper Cu 64 Anti-CEA Monoclonal Antibody M5A PET)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (Copper Cu 64 Anti-CEA Monoclonal Antibody M5A PET) (N=20)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Sinus bradycardia (Cardiac disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, spec (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
General disorders and administration sit (General disorders) | 3 (3)
Catheter related infection (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 15 (15)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT02293954/Prot_SAP_000.pdf